CLINICAL TRIAL: NCT01561469
Title: Multicenter, Retrospective, Observational Study to Evaluate Clinical and Economic Outcomes of Patients With MRSA Hospital-Acquired Pneumonia Treated With Linezolid Or Vancomycin
Brief Title: Evaluation of Patients With Methicillin-Resistant Staphylococcus Aureus Hospital-Acquired Pneumonia Treated With Linezolid or Vancomycin
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: University of Louisville (Other); Henry Ford Hospital (Other); Summa Health System (Other); Sparrow Health System (Other); Jackson Health System (Other)
Responsible Party: Sponsor
Other Study IDs: A5951168
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-06

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus (MRSA); Hospital-Acquired Pneumonia
Keywords: Linezolid; Vancomycin; Ventilator-Associated Pneumonia; Respiratory Tract Infections
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Respiratory Tract Infections | interventions — Linezolid; Vancomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Linezolid observational cohort
  Interventions: Drug: Linezolid
- Vancomycin observational cohort
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Linezolid — Patients with documented MRSA hospital-acquired or ventilator-associated pneumonia treated with linezolid according to routine medical care.
  Other Names: Zyvox
  Groups: Linezolid observational cohort
Drug: Vancomycin — Patients with documented MRSA hospital-acquired or ventilator-associated pneumonia treated with vancomycin according to routine medical care.
  Other Names: Vancocin
  Groups: Vancomycin observational cohort

SUMMARY:
The objective of this study is to review the local management of patients with methicillin-resistant Staphylococcus aureus hospital-acquired pneumonia treated with vancomycin or linezolid with the goal to define if any difference exists among these antimicrobials in regard to clinical and economic outcomes.

DETAILED DESCRIPTION:
Non-randomized, retrospective, observational study

ELIGIBILITY:
Inclusion Criteria:

Patients will be enrolled in the study if they fulfill the following three inclusion criteria:

1. Protocol criteria for HAP/VAP: Criteria for making a correct diagnosis of HAP will be met if the patient develops a new or progressive pulmonary infiltrate associated with at least two of the following: new or increased respiratory symptomatology (cough, sputum or tracheal secretions, shortness of breath), fever or hypothermia, leukocytosis, left shift, or leukopenia, or deterioration of pulmonary function.
2. Isolation of MRSA from a respiratory sample or blood culture within 48 hours of the diagnosis of HAP/VAP
3. Treatment of MRSA HAP/VAP with either vancomycin or linezolid with incorporation of 100 patients in the vancomycin arm and 100 patients in the linezolid arm

Exclusion Criteria:

Patients not meeting enrollment criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This non-interventional study will retrospectively evaluate patients with documented MRSA hospital-acquired including ventilator-associated pneumonia treated with linezolid or vancomycin with incorporation of 100 patients in the vancomycin arm and 100 patients in the linezolid arm.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951168&StudyName=Evaluation%20of%20Patients%20with%20Methicillin-Resistant%20Staphylococcus%20aureus%20Hospital-Acquired%20Pneumonia%20Treated%20with%20Linezolid%20or%20Vancomycin

RESULTS

PARTICIPANT FLOW:
Groups:
- Linezolid: Participants with diagnosis of ventilator-associated pneumonia (VAP) (subgroup of hospital-acquired pneumonia [HAP]) due to methicillin-resistant staphylococcus aureus (MRSA) and who were treated with linezolid according to routine local care were observed retrospectively for up to 28 days after the diagnosis of VAP.
- Vancomycin: Participants with diagnosis of ventilator-associated pneumonia (VAP) (subgroup of hospital-acquired pneumonia [HAP]) due to methicillin-resistant staphylococcus aureus (MRSA) and who were treated with vancomycin according to routine local care were observed retrospectively for up to 28 days after the diagnosis of VAP.
Period: Overall Study
Arm/Group | Linezolid | Vancomycin
Started | 101 | 87
Completed | 101 | 87
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who met the eligibility criteria for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Linezolid | Vancomycin | Total
Number analyzed (Participants) | 101 | 87 | 188
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [48 to 68] | 56 [40 to 66] | 57 [45.75 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 63 | 49 | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Success
Description: Clinical success was assessed as number of participants cured or improved. Cure = complete resolution of signs and symptoms of pneumonia; Improvement = partial resolution of signs and symptoms of pneumonia.
Time Frame: 14 days after diagnosis with VAP or hospital discharge, whichever occurred first
Population: Analysis population included all participants who met the eligibility criteria for this study.
Measure: Number; unit: percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 101 | 87
percentage of participants | 85 | 69
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Test type: Superiority or Other; p = 0.009, Regression, Logistic

2. Secondary Outcome: Number of Participants With Microbiological Outcome
Description: Microbiological outcome was defined as superinfections (infections diagnosed within 72 hours of the diagnosis of HAP and until day 28) and colonization (positive cultures with a multi-drug resistant organism).
Time Frame: 28 days after diagnosis of VAP
Population: Analysis population included all participants who met the eligibility criteria for this study.
Measure: Number; unit: participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 101 | 87
participants
  Superinfections | 42 | 37
  Colonization | 34 | 32
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Analysis for superinfections category reported; Test type: Superiority or Other; p = 1.00, Chi-squared
Statistical Analysis 2: Comparison: Linezolid vs Vancomycin; Analysis for colonization category reported; Test type: Superiority or Other; p = 0.759, Chi-squared

3. Secondary Outcome: Duration of Hospital Stay
Description: Duration of hospital stay was assessed as number of days from VAP diagnosis to discharge from the hospital.
Time Frame: Up to 28 days after diagnosis of VAP
Population: Analysis population included all participants who met the eligibility criteria for this study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 101 | 87
days | 18 [10 to 28] | 16 [11 to 25.5]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Test type: Superiority or Other; p = 0.773, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Description: Duration of ICU stay was assessed as number of days from VAP diagnosis to discharge from the ICU.
Time Frame: Up to 28 days after diagnosis of VAP
Population: Analysis population included all participants who met the eligibility criteria for this study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 101 | 87
days | 11 [8 to 22] | 13 [8 to 19.5]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Test type: Superiority or Other; p = 0.823, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration of mechanical ventilation was assessed as number of days from VAP diagnosis to extubation or to discharge if not extubated.
Time Frame: Up to 28 days after diagnosis of VAP
Population: Analysis population included all participants who met the eligibility criteria for this study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 101 | 87
days | 11 [11 to 24] | 13 [9.5 to 24]
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Test type: Superiority or Other; p = 0.276, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Duration of Antimicrobial Treatment
Time Frame: Up to 28 days after diagnosis of VAP
Population: Analysis population included all participants who met the eligibility criteria for this study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 101 | 87
days | 11 (4) | 11 (5)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Test type: Superiority or Other; p = 0.512, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Antibiotic Free Days
Time Frame: Up to 28 days after diagnosis of VAP
Population: Data was not analyzed for this outcome because other reported measures (that is, duration of antimicrobial treatment, duration of mechanical ventilation, duration of ICU stay, duration of hospital stay) were considered to represent a more strict and useful reflection of resource utilization.
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Due to retrospective nature of the study, adverse events data was not collected.
Arm/Group | Linezolid | Vancomycin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Prioritization of endpoints as primary or secondary was not specified in protocol and was based on study team's inputs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.